CLINICAL TRIAL: NCT06249672
Title: Longterm Functional Outcomes in Patients Undergoing Organ Preserving Treatment for Rectal Cancer With or Without Local Excision After Chemoradiotherapy
Acronym: PRESERVE
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02252
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Organ preservation without local excision
- Organ preservation after local excision
  Interventions: Other: Local excision

INTERVENTIONS:
Other: Local excision — Organ preservation after RCT (radiochemotherapy) of rectal cancer
  Groups: Organ preservation after local excision

SUMMARY:
Treatment of rectal cancer by standard neoadjuvant chemoradiotherapy protocols leads to a complete response in about 15% of patients, or even a higher fraction if radiotherapy is followed by an Oxaliplatin based chemotherapy as published recently.

If patient presents with a (near) complete response at the time of restaging after neoadjuvant treatment, an organ preservation strategy can be an alternative treatment to low anterior resection or abdominoperineal excision of the rectum. An organ preserving strategy is an ideal option for patients that are too frail for a major oncological resection. Furthermore, organ preservation is increasingly an option for a broader spectrum of patients as there is growing evidence that it allows to avoid surgical risks, including major dysfunction of the urinary, sexual and anorectal function at equivalent oncological outcomes.

Studies investigating organ preserving rectal cancer treatment can broadly be divided into two categories. The first option is a planned local resection of the remaining scar at the site of the tumor after chemoradiotherapy. This can be achieved by direct transanal resection in very low tumors or by an endoscopic procedure as TEM (transanal endoscopic microsurgery) or TAMIS (trans-anal minimally invasive surgery). The advantage of this approach is the resulting pathological diagnosis which can confirm the complete response microscopically or indicate if there is remnant tumor tissue left and whether this is completely removed. However, local resection might have an additional negative functional impact and cumulate with function impairment from chemoradiotherapy.

Alternatively, patients after complete clinical response can directly enter a surveillance programme without excision of the remaining scar after neoadjuvant treatment. This strategy provides less certainty about the complete regression of the primary tumor, but allows a treatment completely without surgical interventions and might lead to an even better functional outcome compared to patients undergoing local excision.

There is good evidence that the influence of chemoradiotherapy on anorectal and genitourinary function is relevant. However there is lack of good quality data how much local excision adds to this impairment on the long run. In this study the investigator aims to compare functional outcomes and subjective treatment satisfaction in patients undergoing organ preserving treatment for rectal cancer with and without local resection after chemoradiotherapy. This data will help patients and healthcare personal to choose between these treatment options in the future, knowing the difference in functional outcome between the groups.

As this is an observational study, there will not be any influence on treatment decisions for the included subjects. Clinical data will be collected by questionnaires and compared between the two cohorts, which is in line with a risk category A according to HRO (Human Research Ordinance).

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Informed consent
* Diagnosis of rectal cancer, <12cm from anal verge
* Treatment by chemoradiation (short course 5x5 Gy or 28x1.8 Gy with concomitant 5FU)
* Re staging with MRI/endoscopy shows (near) complete response (max 2cm tumor scar)
* Decision for treatment by organ preservation strategy (with or without local excision)

Exclusion Criteria:

* Inability to give consent
* Follow-up not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for rectal cancer at Bern University hospital have to be discussed in the colorectal MDT per institutional guidelines. In order to identify all eligible patients, MDT lists are screened weekly and all patients meeting in-/exclusion criteria asked for consent. If consent is given, participants will be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Low anterior resection syndrome | 24 months
  LARS (Low Anterior Resection Syndrome) according standardized questionnaire with a range of 0 to 40 points.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kohler, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Bern University Hospital, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No